CLINICAL TRIAL: NCT01934712
Title: A Trial Investigating the Pharmacokinetic Properties of FIAsp in Japanese Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3918; U1111-1121-2896 (Other: WHO); JapicCTI-132253 (Registry Identifier: JAPIC)
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIAsp (Experimental): Each subject will be randomly allocated to one of the two treatment sequences consisting of 2 dosing visits
  Interventions: Drug: Faster-acting insulin aspart; Drug: insulin aspart
- NovoRapid® (Active Comparator): Each subject will be randomly allocated to one of the two treatment sequences consisting of 2 dosing visits
  Interventions: Drug: Faster-acting insulin aspart; Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Single dose injected subcutaneously (s.c, under the skin)
Drug: insulin aspart — Single dose injected subcutaneously (s.c, under the skin)

SUMMARY:
This trial is conducted in Japan. The aim of the trial is to evaluate the pharmacokinetic (the exposure of the trial drug in the body) and pharmacodynamic (the effect of the trial drug on the body) properties of FIAsp (faster-acting insulin aspart) and the currently marketed insulin aspart (NovoRapid®) in Japanese subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for 12 months or longer
* Body mass index (BMI) 18.5-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking at least one cigarette, cigar or pipe daily)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2014-01-28 (Actual); Study Completion 2014-01-28 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0-1 hour

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0-12 hours
Area under the glucose infusion rate (GIR) curve | From 0-1 hour
Area under the glucose infusion rate (GIR) curve | From 0-12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Fukuoka, Japan

REFERENCES:
- [Background] Shiramoto M, Nishida T, Hansen AK, Haahr H. Fast-acting insulin aspart in Japanese patients with type 1 diabetes: Faster onset, higher early exposure and greater early glucose-lowering effect relative to insulin aspart. J Diabetes Investig. 2018 Mar;9(2):303-310. doi: 10.1111/jdi.12697. Epub 2017 Jul 7. PMID 28556616
- [Result] Haahr H, Pieber TR, Mathieu C, Gondolf T, Shiramoto M, Erichsen L, Heise T. Clinical Pharmacology of Fast-Acting Insulin Aspart Versus Insulin Aspart Measured as Free or Total Insulin Aspart and the Relation to Anti-Insulin Aspart Antibody Levels in Subjects with Type 1 Diabetes Mellitus. Clin Pharmacokinet. 2019 May;58(5):639-649. doi: 10.1007/s40262-018-0718-6. PMID 30402720
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com